CLINICAL TRIAL: NCT02318342
Title: Assessment of TRanscathetEr and Surgical Aortic BiOprosthetic Valve Dysfunction With Multimodality Imaging and Its TrEatment With Anticoagulation
Brief Title: Assessment of TRanscathetEr and Surgical Aortic BiOprosthetic Valve Thrombosis and Its TrEatment With Anticoagulation
Acronym: RESOLVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Raj Makkar, Associate Director, Cedars-Sinai Heart Institute; Professor of Medicine, University of California, Los Angeles; Director, Cardiac Catheterization Laboratories and Intervention Center, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSMC-37587
Record Dates: First submitted 2014-12-04; First posted 2014-12-17 (Estimated); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Prosthetic Valve Thrombosis
MeSH Terms: interventions — Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pre-existing bioprosthetic aortic valve (Experimental): Patients with a history of surgical or transcatheter valve replacement with bioprosthetic valves undergo cardiac contrast CT imaging and transthoracic echocardiography to evaluate structural and functional integrity of the aortic valves. Patients with prosthetic valve abnormalities suggestive of thrombus will be administered anticoagulation therapy with Vitamin K antagonists (Warfarin) for 3 months with goal INR 2-3, followed by repeat contrast CT of the chest and transthoracic imaging. Repeat imaging following 3 months of anticoagulation therapy is performed to evaluate the response to anticoagulation therapy.
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Warfarin — Patients with prosthetic valve abnormalities suggestive of thrombus will be administered anticoagulation therapy with Vitamin K antagonists (Warfarin) for 3 months with goal INR 2-3, followed by repeat contrast CT of the chest and transthoracic imaging. Repeat imaging following 3 months of anticoagulation therapy is performed to evaluate the response to anticoagulation therapy.
  Other Names: Coumadin

SUMMARY:
This is a prospective study designed to evaluate the structural and functional integrity of transcatheter or surgical bioprosthetic valves with multimodality imaging. The study further aims to confirm resolution of the early bioprosthetic valve thrombotic changes with anticoagulation.

DETAILED DESCRIPTION:
Patients with a history of bioprosthetic valve replacement undergo cardiac contrast CT imaging and transthoracic echocardiography to evaluate structural and functional integrity of the aortic valves. The imaging studies will be performed at least 48-hours after bioprosthetic valve replacement. Patients with prosthetic valve abnormalities suggestive of thrombus will be administered anticoagulation therapy, followed by repeat contrast CT of the chest and transthoracic imaging. Repeat imaging following 3 months of anticoagulation therapy is performed to evaluate the response to anticoagulation therapy. I

ELIGIBILITY:
Inclusion Criteria:

* Presence of transcatheter or surgical bioprosthetic aortic valve implanted at least 48 hours prior to enrollment
* Age 18 years or older
* Ability to provide informed consent and follow-up with protocol procedures.

Exclusion Criteria:

* Renal insufficiency (creatinine > 1.5 mg/dL)
* Known allergy to iodinated contrast agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2014-12; Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of patients with structural/functional abnormalities of bioprosthetic valves | 3 months

OTHER OUTCOMES:
Percentage of patients with resolution of bioprosthetic valve thrombotic lesions with anticoagulation | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Raj Makkar, MD, Principal Investigator — Cedars-Sinai Medical Center, Los Angeles, California
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Makkar RR, Fontana G, Jilaihawi H, Chakravarty T, Kofoed KF, De Backer O, Asch FM, Ruiz CE, Olsen NT, Trento A, Friedman J, Berman D, Cheng W, Kashif M, Jelnin V, Kliger CA, Guo H, Pichard AD, Weissman NJ, Kapadia S, Manasse E, Bhatt DL, Leon MB, Sondergaard L. Possible Subclinical Leaflet Thrombosis in Bioprosthetic Aortic Valves. N Engl J Med. 2015 Nov 19;373(21):2015-24. doi: 10.1056/NEJMoa1509233. Epub 2015 Oct 5. PMID 26436963
- [Background] Chakravarty T, Sondergaard L, Friedman J, De Backer O, Berman D, Kofoed KF, Jilaihawi H, Shiota T, Abramowitz Y, Jorgensen TH, Rami T, Israr S, Fontana G, de Knegt M, Fuchs A, Lyden P, Trento A, Bhatt DL, Leon MB, Makkar RR; RESOLVE; SAVORY Investigators. Subclinical leaflet thrombosis in surgical and transcatheter bioprosthetic aortic valves: an observational study. Lancet. 2017 Jun 17;389(10087):2383-2392. doi: 10.1016/S0140-6736(17)30757-2. Epub 2017 Mar 19. PMID 28330690
- [Derived] Nagasaka T, Patel V, Suruga K, Guo Y, Koren O, Shechter A, Friedman M, Patel D, Chakravarty T, Cheng W, Gupta A, Ishii H, Jilaihawi H, Nakamura M, Makkar RR. Prognostic implications and predictive factors of subclinical leaflet thrombosis following valve-in-valve transcatheter aortic valve implantation. EuroIntervention. 2025 May 5;21(9):e482-e492. doi: 10.4244/EIJ-D-24-00711. PMID 40325986
- [Derived] Nagasaka T, Patel V, Shechter A, Suruga K, Koren O, Chakravarty T, Cheng W, Ishii H, Jilaihawi H, Nakamura M, Makkar RR. Impact of Balloon-Expandable TAVR Valve Deformation and Calcium Distribution on Outcomes in Bicuspid Aortic Valve. JACC Cardiovasc Interv. 2024 Sep 9;17(17):2023-2037. doi: 10.1016/j.jcin.2024.07.018. PMID 39260960
- [Derived] Raschpichler M, Flint N, Yoon SH, Kaewkes D, Patel C, Singh C, Patel V, Kashif M, Borger MA, Chakravarty T, Makkar R. Commissural Alignment After Balloon-Expandable Transcatheter Aortic Valve Replacement Is Associated With Improved Hemodynamic Outcomes. JACC Cardiovasc Interv. 2022 Jun 13;15(11):1126-1136. doi: 10.1016/j.jcin.2022.04.006. PMID 35680192
- [Derived] Ochiai T, Oakley L, Sekhon N, Komatsu I, Flint N, Kaewkes D, Yoon SH, Raschpichler M, Patel V, Tiwana R, Enta Y, Mahani S, Kim Y, Stegic J, Chakravarty T, Nakamura M, Cheng W, Makkar R. Risk of Coronary Obstruction Due to Sinus Sequestration in Redo Transcatheter Aortic Valve Replacement. JACC Cardiovasc Interv. 2020 Nov 23;13(22):2617-2627. doi: 10.1016/j.jcin.2020.09.022. PMID 33213747
- [Derived] Ochiai T, Chakravarty T, Yoon SH, Kaewkes D, Flint N, Patel V, Mahani S, Tiwana R, Sekhon N, Nakamura M, Cheng W, Makkar R. Coronary Access After TAVR. JACC Cardiovasc Interv. 2020 Mar 23;13(6):693-705. doi: 10.1016/j.jcin.2020.01.216. PMID 32192689